CLINICAL TRIAL: NCT01026259
Title: Local Warming: Effects on Wound Infection and Healing
Brief Title: Local Warming of Surgical Incisions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: JoAnne Whitney, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 29991-A
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Surgical Wound Infection
Keywords: Surgical site infection; wound healing; tissue oxygen; angiogenesis; flow cytometry; immunohistochemistry
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local incision warming (Experimental): Local warming applied to surgical incision for 6 treatments beginning in post anesthesia recovery through the second postoperative day.
  Interventions: Other: Warming of surgical incision
- No warming to surgical incision (Active Comparator): Incisions covered with same postoperative dressing as in Arm 1 but without warming treatments.
  Interventions: Other: Warming dressing without actual warming

INTERVENTIONS:
Other: Warming of surgical incision — A warming pack (chemical activation) is applied to the dressing over the surgical incision, warming to 38 degrees C, for a period of 90 minutes times 6 treatments. The first treatment occurs in the PACU.
  Arms: Local incision warming
Other: Warming dressing without actual warming — The same type of surgical incision dressing is used but no warming treatments are administered.
  Arms: No warming to surgical incision

SUMMARY:
The purpose of this study is to determine if local warming of surgical wounds improves healing and helps prevent infection. The investigators want to see if warming surgical incisions improves oxygen levels and healing in skin close to the incision.

DETAILED DESCRIPTION:
Surgical site infections (SSI) account for 37% of US hospital infections and increase morbidity and cost. High rates (10-22%) of SSI are associated with colorectal surgery and obesity. Bacterial resistance requires oxygen and higher tissue oxygen limits infection in general surgery patients. Control of core and local temperature may increase infection resistance by modulating perfusion, oxygenation, angiogenesis and immune cell responses. Perioperative hypothermia reduces tissue oxygen while normothermia lowers SSI rates. Warming injured tissues locally may offer additional benefit. Warming incisions immediately after surgery and intermittently for two days after gastric bypass or colectomy surgery reduced infection rates in a pilot sample. Systematic study of clinical outcomes and potential mechanisms in a larger study is lacking and is the focus of the current study.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older,
* scheduled for bariatric, colon or gynecological surgery,
* able to speak and read English.

Exclusion Criteria:

* glucocorticoids greater than 5 mg per day,
* albumin below 3.0,
* creatinine above 2.5 mg/dl,
* history of pulmonary edema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2005-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | Within 6 weeks of the surgical procedure

SECONDARY OUTCOMES:
Wound tissue response | First 9 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States